CLINICAL TRIAL: NCT05600634
Title: Multi Center Clinical Observation of Sentinel Skin Graft From the Same Donor Source for Detecting Acute Rejection After Renal Transplantation
Brief Title: Multi Center Observation of Sentinel Skin Graft for Detecting Acute Rejection After Renal Transplantation
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0719
Record Dates: First submitted 2022-10-27; First posted 2022-10-31 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant Rejection; Skin Graft

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney and skin transplataiton
  Interventions: Procedure: Skin allotransplantation

INTERVENTIONS:
Procedure: Skin allotransplantation — Sentinel skin grafts from the same donor source will be carried on in the meantime of kidney transplantation for assisting to detect acute renal rejection.

SUMMARY:
The purpose of this study was to explore the accuracy of sentinel skin grafts from the same donor source in diagnosing renal allograft rejection, and to provide new ideas and options for the later clinical diagnosis of renal allograft rejection. Further, try to provide timing guidance for early immunization intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end-stage renal disease undergoing renal transplantation;
2. 18-60 years old;
3. Postoperative follow-up points are complete (visit the hospital every week in the first month after surgery, every two weeks in 2-3 months, every four to six months, and every three months in 7-12 months. Follow up at any time when skin rejection is observed. The follow-up time may be adjusted when the condition changes);
4. The participants had good compliance, volunteered to participate in the test and signed the informed consent form.

Exclusion Criteria:

1. Untreated or disseminated malignant tumor;
2. Active period of infectious diseases;
3. Serious cardiovascular disease occurred recently;
4. Combined with other important organ failure;
5. History of mental illness or cognitive impairment;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study is an exploratory study. In the early stage, there is no relevant study on the accuracy of sentinel skin flap monitoring renal rejection, and there is a lack of corresponding sensitivity and specificity indicators. Considering that the incidence of acute rejection in the first year after transplantation is 15-30%, it is estimated that 20 cases will be included. Because the experimental data may be lost, or the participants may withdraw from the trial or lose the interview, the sample size will be increased by 20%, and finally 24 cases will be included in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2017 Banff Kidney Transplantation Rejection Rating | Through study completion, an average of 1 year
  A rating evaluation on kidney rejection
2007-edition Banff skin containing allogeneic composite histopathological diagnosis grading | Through study completion, an average of 1 year
  Skin histopathological diagnosis
Renal function testing | Through study completion, an average of 1 year
  Blood Cr and Bun testing

SECONDARY OUTCOMES:
Renal ultrasound diagnosis | Through study completion, an average of 1 year
  Renal ultrasound diagnosis
Complications | Through study completion, an average of 1 year
  Complications assessment

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Xijing Hospital, Ari Force Medical University, Xi'an, Shannxi
  - First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No